CLINICAL TRIAL: NCT00724256
Title: Randomised Controlled Trial on Efficacy and Safety of Short Term Versus Long Term Antibiotic Therapy for Pyelonephritis in Childhood.
Brief Title: Short-term Antibiotic Therapy for Pyelonephritis in Childhood
Acronym: STUTI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: other upcoming studies; patients refusal of invasive follow up (DMSA)
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Marzia Lazzerini, MD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTI_62-2006
Record Dates: First submitted 2008-07-18; First posted 2008-07-29 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Pyelonephritis
Keywords: Pyelonephritis.; Urinary Tract Infections.; Children.; Randomised controlled trial.; Therapy.; Ceftibuten.
MeSH Terms: conditions — Pyelonephritis; Urinary Tract Infections | interventions — Ceftibuten

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ceftibuten
- 2 (Active Comparator)
  Interventions: Drug: ceftibuten

INTERVENTIONS:
Drug: ceftibuten — ceftibuten 9mg/kg once a day for 7 days.
  Arms: 1
Drug: ceftibuten — ceftibuten 9mg/kg once a day for 10 days.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of oral ceftibuten for 7 days versus 10 days in acute pyelonephritis in children.

The main hypothesis is that the ceftibuten for 7 days will be not inferior to ceftibuten 10 days in the rate of renal scarring at 6-12 months.

DETAILED DESCRIPTION:
Acute pyelonephritis is one of the most common serious bacterial infections in childhood, particularly in young children, with an estimated prevalence in febrile infants of 5.3%. It has been considered an important risk factor for the development of renal scarring, and renal insufficiency. More recently the long term outcomes of pyelonephritis has ameliorated, probably because of prompt diagnosis and therapy, and the importance of urinary tract infection as a risk factor for renal insufficiency has been questioned.

Nevertheless, the optimal type and duration of antibiotic therapy for acute uncomplicated pyelonephritis in children is not established yet.

There is a general agreement that children who are dehydrated, unable to drink, or in whom sepsis is possible, should be admitted to hospital for intravenous antibiotic treatment.

Outside this conditions, evidence suggest that children with acute pyelonephritis can be treated effectively with cefixime, ceftibuten or amoxycillin/clavulanic acid. given orally (1).

A recently updated Cochrane review on antibiotic treatment for acute pyelonephritis in children identified twenty three studies (3407 children). No significant differences were found in persistent renal damage at six to 12 months (824 children: RR 0.80, 95% CI 0.50 to 1.26) or in duration of fever (808 children: WMD 2.05, 95% CI -0.84 to 4.94) between oral antibiotic therapy (10 to 14 days) and IV therapy (3 days) followed by oral therapy (10 days). Similarly no significant differences in persistent renal damage (3 studies, 341 children: RR 1.13, 95% CI 0.86 to 1.49) were found between IV therapy (3 to 4 days) followed by oral therapy and IV therapy for 7 to 14 days.

Authors concluded that children with acute pyelonephritis can be treated effectively with oral antibiotics (cefixime, ceftibuten and amoxycillin/clavulanic acid) or with short courses (2 to 4 days) of IV therapy followed by oral therapy.

Oral treatment also is easier to use and does not require admission to hospital, leading to reduced costs.

Nevertheless, the exact duration of oral therapy is not established. Current guidelines recommend 7-14 days course of broad-spectrum antibiotics capable of reaching significant renal levels.

The objective of our study is to evaluate if oral ceftibuten for 7 days is equally effective as oral ceftibuten for 10 days in acute pyelonephritis in children.

This is a non-inferiority randomised controlled trial to determine whether a short term therapy with ceftibuten ( 7 days) will be therapeutically similar to a long term therapy ( 10 days), measuring as major outcome the prevalence of renal scars.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 5 years, with a first episode of pyelonephritis.

Exclusion Criteria:

* Children less than 1 month, or older than 5 years.
* Relapse of pyelonephritis.
* Sepsis and/or vomiting, or other conditions where it's impossible to administer an oral therapy.
* Allergy to ceftibuten.
* Previous antibiotic therapy for the same infection.
* Long term antibiotic prophylaxis with an antibiotic of the same class, if laboratory antibiotic resistance is shown.
* Children with uncontrolled other disease.
* Complicated pyelonephritis (abscess).

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Rate of renal SCAR | 6-12 month from urinary tract infection

SECONDARY OUTCOMES:
Relapses | up to12 months
Adverse effects of drug therapy | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Lazzerini, MD DTMH, Study Director — IRCCS Burlo Garofolo
Locations (1):
- Institute for Child Health Burlo Garofolo, Trieste, Triest, Italy

REFERENCES:
- [Background] Hodson EM, Willis NS, Craig JC. Antibiotics for acute pyelonephritis in children. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003772. doi: 10.1002/14651858.CD003772.pub3. PMID 17943796